CLINICAL TRIAL: NCT01736046
Title: Effects of CT Reconstruction Algorithm on the Quantitative Assessment of Crohn's Disease: A Comparison of Standard and Low Dose CT Enterography
Brief Title: Comparison of Standard and Low Dose CT Enterography for Crohn's Disease
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H12-02211
Record Dates: First submitted 2012-11-06; First posted 2012-11-29 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Crohn's Disease
Keywords: CT Enterography; Crohn's Disease; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Crohn's Disease patients: All patients referred for CT Enterography will be undergo both standard and low dose CT Enterography
  Interventions: Radiation: CT Enterography

INTERVENTIONS:
Radiation: CT Enterography — Diagnostic CT Enterography Scan (CTE)
  Subjects will have their scheduled diagnostic CTE scan done according to St. Paul's Hospital radiology department standard procedures. Subjects will be randomly assigned to undergo a low dose CT Enterography scan either before or after the diagnostic scan. The radiologists who are blinded to the technique used will then interpret the scans to look for signs of Crohn's disease. The low dose scan will be compared to the standard scan in terms of it's ability to detect signs of Crohn's disease.
  Other Names: CT Scan to include imaging of the small bowel and colon

SUMMARY:
The investigators will be assessing the efficacy of a Model Based Iterative Reconstruction algorithm (MBIR) as a noise reduction tool in computed tomographic (CT) examinations for Crohn's Disease. MBIR is computer adapted mathematical calculation technique that generates CT images with less picture degradation (noise) than traditional computer reconstruction techniques such as FBP (Filtered Back Projection) and ASIR (Adaptive Statistical Iterative Reconstruction), for enteric Crohn's Disease findings.

The research involves collection of data from subjects standard of care diagnostic CT scan and from a research low radiation dose scan performed immediately following their diagnostic scan. We will determine the impact on image quality, interpretability, and Crohn's Disease findings of the low dose scan compared to the standard of care scan.

FBP, MBIR, and ASIR are post processing tools that do not alter the scan acquisition itself.

DETAILED DESCRIPTION:
1. PURPOSE

   The purpose of this study is to assess the efficacy of a new model based iterative reconstruction algorithm as a noise reduction tool and to compare its sensitivity for the findings of enteric Crohn's Disease with the sensitivity of FBP or ASIR CT Enterography findings in enteric Crohn's Disease.

   Definitions:

   Iterative reconstruction: A computer adapted mathematical calculation technique that allows the ability to generate CT images with less image noise (picture degradation) than traditional image reconstruction techniques.

   Reconstruction algorithms are computer adapted mathematical calculations applied to raw data during image reconstruction.
2. HYPOTHESIS

   The use of different CT reconstruction algorithms will allow the quantitative assessment of small bowel Crohn's Disease (CD) while exposing patients to lower radiation doses. MBIR and ASIR will provide images with lower noise and similarly accurate quantification of CD. Additionally, MBIR will allow acquisition of CT data at very low radiation doses, with comparable image quality and quantitative assessment of CD compared to higher radiation dose acquisitions performed utilizing FBP and ASIR. MBIR will not be inferior to FBP or ASIR in assessing findings related to Crohn's Disease on CT enterography (CTE).

   Definitions

   MBIR: Model Based Iterative Reconstruction algorithm FBP: Filtered Back Projection ASIR: Adaptive Statistical Iterative Reconstruction
3. JUSTIFICATION

   Computed tomography imaging traditionally relied upon filtered back projection (FBP) for image reconstruction. This technique uses relatively little computing power, but requires a number of assumptions be made about the data acquisition itself that result in an increase in image noise.

   The use of iterative reconstruction techniques has recently started to take place in CT imaging. The major benefit of iterative reconstruction techniques is the ability to generate CT images with less image noise. This noise reduction allows for tube current reduction with IR images, limiting radiation dose in a linear manner.

   Model based iterative reconstruction (MBIR), is replacing the older iterative technique, adaptive statistical iterative reconstruction (ASIR). MBIR utilizes more accurate modeling and early research suggests MBIR images may be reconstructed from CT acquisitions that use significantly decreased radiation dose, with similar image quality compared to both ASIR and FBP.

   FBP, MBIR, and ASIR are post processing tools that do not alter the scan acquisition itself. Iterative reconstruction algorithms have garnered increased interest, especially with elevated public concern about radiation dose . MBIR techniques have not yet been validated in CT examinations acquired for evaluation of Crohn's Disease (CD).

   Clinical history, physical examination, laboratory investigations and endoscopy have been used to identify and evaluate the extent and severity of Crohn's Disease along with imaging studies to assist in the evaluation of the small bowel involvement of CD. CT Enterography has become the preferred imaging modality for assessing small bowel involvement in inflammatory bowel disease. The dose reduction properties of MBIR are particularly appealing in this area of CT imaging as multiple scans may be performed over time to assess progression or relapse of disease and response to treatment.

   Calprotectin is a protein found inside the cytoplasm of the immune cells within the intestine known as neutrophils, granulocytes and macrophages. Under conditions of mucosal inflammation as seen in inflammatory bowel disease, calprotectin is released into the lumen of the bowel and excreted in the stool. Fecal Calprotectin levels can be measured and serve as a biological marker of the degree of mucosal inflammation in the bowel. Fecal calprotectin levels have not been previously correlated with the degree of mucosal inflammation seen on CT Enterography.
4. OBJECTIVE

   To determine the impact on image quality, interpretability, and Crohn's Disease findings of low dose computed tomography enterography (CTE) images acquired with a new model based iterative reconstruction algorithm as compared to standard image reconstruction.
5. RESEARCH METHOD

   The research is a prospective non randomized study of 163 consecutive patients who are clinically referred for CT Enterography.
6. STATISTICAL ANALYSIS

Using sensitivity of the CTE to calculate sample size, the planned sample size for this study is 163 subjects. The study will be powered at 80% to demonstrate that the lower radiation CTE (ASIR and MBIR) is non-inferior (type I error rate of 2.5%, one sided) to the standard CTE. The sensitivity of the standard CTE is assumed to be 0.77 based on a pooled estimate [7]. 0.1 is chosen as the non-inferiority margin. The correlation between the two procedures is considered in the sample size calculation. We assume that the prevalence of Crohn's Disease is 80% among the target population.

Using the nQuery statistical program, with the assumption that the proportion of discordant examinations is 0.15(or the conditional probability of positive finding in standard CTE is 0.90 if given a positive finding on the ASIR or MBIR CTE), the sample size needed to detect no more than 0.1 difference in sensitivity of the two procedures for patients with disease is 118, with a 80% power and a type I error of 0.025, one sided. Assuming that 80% of target population will have disease, approximately 148 subjects will need to be recruited. We have factored in a 10% drop out rate ( patients who leave the study for any reason) bringing the total number of patients to be recruited to 163.

Image quality scores and quantitative analysis will be compared using both standard and the novel reconstruction algorithms. These results will also be compared to the acquired FC levels. Because each patient examination will receive multiple reconstructions, a mixed-model analysis will be conducted to account for repeated observations within patients. Repeated measures analysis of variance will be conducted separately for each outcome (signal, noise, SNR, proportion of interpretable segments, and image quality) against the type of reconstruction used. A 0.05 significance level will be used for all repeated measures and analysis.

Primary Endpoint:

FBP, ASIR and MBIR will each be compared to the reference standard described below. The endpoint will be the ability of each method to accurately identify the presence or absence of Crohn's Disease (CD) as compared to the reference standard.

Reference Standard:

Dr. B. Bressler, the principal investigator, is a gastroenterologist with an expertise in inflammatory bowel disease (IBD). Dr. Bressler will review all of the available clinical parameters including history and physical exam findings, ileocolonoscopy findings if available and laboratory parameters including bloodwork and Fecal Calprotectin levels. The gastroenterologist will not be blinded to the subject's identity. Based on his review of the above parameters, he will rate the presence of small bowel CD as definitely active, probably active, inactive (remission) or absent.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 19 years or older with suspected or known inflammatory bowel disease referred to the St. Paul's Hospital Radiology department for CT Enterography examination will be eligible to participate.

Exclusion Criteria:

* Patients unable to tolerate oral contrast media ( PegLyte (polyethylene glycol) for bowel distension or with kidney disease (gfr<60) where intravenous contrast would be contraindicated.
* Patients with a known or suspected allergy/reaction to contrast material.
* Pregnant patients Note: As per standard of care in the SPH radiology department, a screening pregnancy test will be done if the patient is of child bearing potential and is not sure that they are pregnant.
* Patients who are unwilling to sign the consent form will not be eligible for participation.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of having Crohn's Disease who are referred for CT Enterography examination by their gastroenterologist
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Low Dose and Standard dose CTE for detecting active Crohn's Disease | 1 year
  FBP, ASIR and MBIR will each be compared to the reference standard. The endpoint will be the ability of each method to accurately identify the presence or absence of Crohn's Disease (CD) as compared to the reference standard.

SECONDARY OUTCOMES:
Correlation of Fecal Calprotectin with Radiology findings of Crohn's Disease | 1 year
  Fecal Calprotectin levels will be measured and the results will be correlated with findings suggestive of Crohn's Disease on CT Enterography

CONTACTS AND LOCATIONS:
Overall Officials: Brian Bressler, MD, Principal Investigator — UBC
Locations (1):
- St. Paul's Hospital, Vancovuer, British Columbia, Canada